CLINICAL TRIAL: NCT03090347
Title: The Effect of Short-term Overconsumption of Specific Dietary Nutrients on Liver and Adipose Tissue Metabolism
Brief Title: Effects of Dietary Nutrients on Liver and Adipose Tissue Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Oxlip-2017-BBSRC/BHF
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-04

CONDITIONS: NAFLD; Nutrient; Excess
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-sugar diet (Experimental): Participants will be asked to consume a relatively low-fat, high-carbohydrate eucaloric diet enriched in free-sugars (20% total energy).
  Interventions: Other: Overconsumption of specific dietary nutrient

INTERVENTIONS:
Other: Overconsumption of specific dietary nutrient — Subjects will be studied before and then after the consumption of a diet where specific nutrients are provided in excess.

SUMMARY:
In health,adipose tissue stores fat from the diet. If the fat tissue stops storing dietary fat then this increases the chance of it being stored in the liver, which is related to increased risk of heart disease and type 2 diabetes. It has been suggested that having a diet high in sugars or certain fats, may cause the fat tissue and liver to change how they function; we would like to investigate this in detail.

DETAILED DESCRIPTION:
This research aims to investigate how the overconsumption of specific macronutrients may effect adipose tissue and liver metabolism and function. Liver and heart fat content and adipose tissue and liver metabolism fasting and postprandial lipid metabolism will be assessed before and after the specific dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged ≥18 or ≤65 years.
* Body Mass Index ≥19 ≤35 kg/m2
* No medical condition or relevant drug therapy known to affect liver or adipose tissue metabolism.
* Weight stable for the previous 3 months

Exclusion Criteria:

* Patient is unwilling or unable to give informed consent for participation in the study
* A blood haemoglobin <135mg/dL for men and <120mg/dL for women
* Donated (or lost) ≥250 ml of blood in the previous two months.
* On a weight loss diet or have decreased their body weight by >5% in the previous 3 months.
* Have increased their body weight by >5% in the previous 3 months.
* Any metabolic condition or relevant drug therapy
* Current smoker
* History of alcoholism or a greater than recommended alcohol intake (>30 g of alcohol daily for men and >20 g of alcohol daily for women)
* Haemorrhagic disorders
* Anticoagulant treatment
* History of albumin allergy
* Pregnant or nursing mothers
* Women who are taking any contraceptive agent or device including oral contraceptives, hormone replacement therapy (HRT) or who have used these within the last 12 months
* History of severe claustrophobia
* Presence of metallic implants, pacemaker, or are unwilling to remove any piercings
* History of an eating disorder or any other psychological condition that may affect the participants ability to adhere to study intervention/experimental diets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Liver de novo lipogenesis | Within 21 days after starting the intervention diet
  Investigators will utilise stable isotope tracer methodology to measure the change in the contribution of newly synthesised fatty acids to very low density lipoprotein triglyceride

SECONDARY OUTCOMES:
Adipose tissue metabolism | Within 21 days after starting the intervention diet
  Investigators will measure the change in the expression of key lipogenic genes in subcutaneous adipose tissue
Liver fat accumulation | Within 21 days after starting the intervention diet
  Investigators will measure the change in the amount of fat within the liver using MRI/S

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the study, all individual data obtained from participants may potentially be shared with other researchers, both here in the United Kingdom and abroad, in appropriate circumstances. If data is to be shared with other researchers, it will be done so under fully anonymised conditions.